CLINICAL TRIAL: NCT07368283
Title: A Single-arm Phase II Non-inferiority Clinical Study of Limited Target Volume Radiotherapy After Glioblastoma Surgery
Brief Title: Limited Target Volume Radiotherapy After Glioblastoma Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhiping Chen, Director of the Head and Neck Radiation Therapy Department，Jiangxi cancer Hospital, Jiangxi Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025ky249
Record Dates: First submitted 2026-01-06; First posted 2026-01-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma (GBM)
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- limited-field radiotherapy Group (Other)
  Interventions: Radiation: limited-field radiotherapy

INTERVENTIONS:
Radiation: limited-field radiotherapy — limited-field radiotherapy + Concurrent and adjuvant TMZ chemotherapy

SUMMARY:
Research on radiotherapy target volumes for glioblastoma is increasingly focused on exploring more limited yet effective irradiation fields, aiming to achieve local control while minimizing acute and long-term neurotoxicity. Previous retrospective analysis by investigators revealed that local recurrences of glioblastoma are predominantly confined to a narrow margin around the original lesion: 98.3% of recurrences occurred within 0.5 cm of the original T2-FLAIR abnormality, 94.8% within 1 cm of the original T1-enhanced region. These findings have been cited in the ESTRO-EANO treatment guidelines. Building on this evidence, investigators plan to conduct a single-arm, phase II clinical trial to systematically evaluate the efficacy and safety of a 1 cm radiotherapy target volume in post-operative glioblastoma patients.Eligible patients with glioblastoma who have undergone surgical resection will be selected to receive limited-field radiotherapy. The target volume will be defined based on the postoperative MRI enhancing lesion: a 1 cm margin will be added to form the clinical target volume (CTV), followed by a further 0.3 cm margin to create the planning target volume (PTV). A total dose of 60 Gy will be delivered in 30 fractions (2 Gy per fraction, 5 fractions per week). Concurrent and adjuvant chemotherapy will be administered per standard guidelines. The primary efficacy endpoints are the 6-month progression-free survival rate and the incidence of symptomatic radiation-induced brain necrosis of grade 3 or higher. Secondary endpoints include overall survival, patterns of recurrence, neurocognitive function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 years.
* Diagnosed with glioblastoma by surgical pathology, with the extent of resection achieving maximal safe resection.
* Within 2 to 6 weeks after surgery
* In good physical condition with a Karnofsky Performance Status (KPS) score ≥ 60.
* Hematological, hepatic, and renal functions are essentially normal.
* Signed informed consent, willing to undergo treatment and follow-up as stipulated in the study protocol.

Exclusion Criteria:

* Prior history of cranial radiotherapy or other malignant tumors.
* Severe dysfunction of vital organs (e.g., heart, liver, kidneys) that precludes tolerance to radiotherapy.
* Active infection, immune system disorders, or other serious chronic diseases.
* Pregnancy or lactation.
* Psychiatric disorders or severe cognitive impairment that compromises the ability to cooperate with treatment and follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
6m PFS | up to 6 month
  6-month progression-free survival rate
incidence of symptomatic radiation-induced brain necrosis of grade 3 or higher | Up to 24 months

SECONDARY OUTCOMES:
OS | Up to 24 months
  overall survival
Location of first recurrence relative to radiation field (in-field, marginal, or distant) | Up to 24 months
  The spatial relationship between the first documented site of disease recurrence/progression and the original radiation treatment plan will be determined by a core imaging laboratory. Recurrent lesions will be co-registered with the original planning CT/MRI and radiation dose distribution.
  Classification is based on the volume of the recurrent lesion covered by the 95% isodose line of the original prescription dose:
  In-field recurrence: >80% of the recurrent lesion's volume is within the 95% isodose line.
  Marginal recurrence: 20% to 80% of the recurrent lesion's volume is within the 95% isodose line.
  Distant recurrence: <20% of the recurrent lesion's volume is within the 95% isodose line.
  This classification criteria is adapted from the dosimetric analysis methods commonly used in radiotherapy studies (e.g., Patterns offailure for glioblastoma multiforme following limited-margin radiation and concurrent temozolomide. Radiation oncology 2014, 9:130.)
Cognitive function assessed by Mini-Mental State Examination (MMSE) score | Up to 24 months
  Cognitive function assessed by the Mini-Mental State Examination (MMSE). Scores range from 0 to 30, with higher scores indicating better cognitive function.
Cognitive function assessed by Montreal Cognitive Assessment (MoCA) score | Up to 24 months.
  Cognitive function assessed by the Montreal Cognitive Assessment (MoCA). Scores range from 0 to 30, with higher scores indicating better cognitive function.
Health-Related Quality of Life as assessed by the EORTC QLQ-C30 Global Health Status / QoL scale | Up to 24 months
  Score on the Global Health Status / Quality of Life scale (Items 29 & 30) of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). Scale range: 0-100. A higher score indicates a better overall quality of life.
Disease-Specific Quality of Life as assessed by the EORTC QLQ-BN20 summary score | Up to 24 months
  Summary score of the European Organization for Research and Treatment of Cancer Brain Cancer Module (EORTC QLQ-BN20). This scale assesses symptoms and issues specific to brain tumor patients (e.g., future uncertainty, visual disorder, motor dysfunction). Scale range and interpretation should be specified
Quality of Life as assessed by the FACT-Br Total Score | Up to 24 months
  Total score of the Functional Assessment of Cancer Therapy - Brain (FACT-Br). This questionnaire assesses physical, social, emotional, functional well-being, and additional concerns specific to brain tumor patients. Scale range: 0-200. A higher score indicates better quality of life.

IPD SHARING:
Plan to Share IPD: Undecided